CLINICAL TRIAL: NCT03059225
Title: Synchronous rTMS and Computer-integrated Speech Training Applied in Aphasic Patients
Brief Title: rTMS in Aphasic Patients With Neuroimage Assessments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Principal investigator, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-05-003A
Record Dates: First submitted 2017-01-16; First posted 2017-02-23 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Stroke; Aphasia
Keywords: Stroke; Aphasia; rTMS; Functional MRI; Speech training
MeSH Terms: conditions — Stroke; Aphasia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): repetitive transcranial magnetic stimulation (rTMS) intervention of contralesional 1Hz-rTMS for 10 daily sessions.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Sham stimulation (Sham Comparator): Sham treatment for 2-week inhibitory non-dominate hemisphere rTMS program.
  Interventions: Device: Sham stimulation
- High frequency rTMS (Experimental): High-frequency rTMS to ipsilesional region for 10 daily sessions.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — undergo contralesional 1Hz repetitive transcranial magnetic stimulation(rTMS) or high frequency ipsilesional rTMS for 10 daily sessions
  Arms: Experimental; High frequency rTMS
Device: Sham stimulation — 2-week inhibitory non-dominate hemisphere rTMS program
  Arms: Sham stimulation

SUMMARY:
The refinement of repetitive transcranial magnetic stimulation (rTMS) has highlighted its merit in terms of learning programs as a treatment for aftereffect augmentation. Nevertheless, the efficacy of synchronous rTMS protocol integrated with computer-integrated speech training is not well understood. It is also not clear regarding the efficacy of compound bi-hemispheric stimulation protocol. The aim of the study is to investigate language response to these new strategies and to determine the longevity of the therapeutic outcome. Advanced MR neuroimaging techniques, such as fMRI and DTI, are powerful tools to evaluate the concomitant nervous changes after rTMS treatment on aphasic patients. The knowledge from fMRI and DTI microstructural evolution provides insight into underlined mechanism operating the language improvement.

DETAILED DESCRIPTION:
The efficacy of synchronous rTMS protocol integrated with computer-integrated speech training is not well understood. It is also not clear regarding the efficacy of inhibitory or excitatory stimulation protocol. The aim of the study is to investigate language response to these new strategies and to determine the longevity of the therapeutic outcome. Advanced MR neuroimaging techniques, such as fMRI and DTI, are powerful tools to evaluate the concomitant nervous changes after rTMS treatment on aphasic patients. The knowledge from fMRI and DTI microstructural evolution provides insight into underlined mechanism operating the language improvement

ELIGIBILITY:
Inclusion Criteria:

* Aphasic stroke in chronic stage (over 3 months)

Exclusion Criteria:

* No seizure history, no brain surgery history, no electronic device in brain or chest, no dementia

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-02-18 (Actual); Primary Completion 2021-12-23 (Estimated); Study Completion 2021-12-23 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in aphasia level on the Concise Chinese Aphasia Test (CCAT) at 2 Weeks | Up to 12 weeks
  linguistic function assessment

SECONDARY OUTCOMES:
Change from Baseline in the concomitant nervous status on the Functional magnetic resonance imaging (fMRI) at 2 weeks | Up to 12 weeks
  brain activity change in fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yi Tsai, MD, Principal Investigator — Department of physical medicine and rehabilitation, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsai PY, Wang CP, Ko JS, Chung YM, Chang YW, Wang JX. The persistent and broadly modulating effect of inhibitory rTMS in nonfluent aphasic patients: a sham-controlled, double-blind study. Neurorehabil Neural Repair. 2014 Oct;28(8):779-87. doi: 10.1177/1545968314522710. Epub 2014 Feb 13. PMID 24526709
- [Derived] Chou TY, Wang JC, Lin MY, Tsai PY. Low-Frequency vs. Theta Burst Transcranial Magnetic Stimulation for the Treatment of Chronic Non-fluent Aphasia in Stroke: A Proof-of-Concept Study. Front Aging Neurosci. 2022 Jan 14;13:800377. doi: 10.3389/fnagi.2021.800377. eCollection 2021. PMID 35095477
- [Derived] Lee IT, Huang CC, Hsu PC, Lin CP, Tsai PY. Resting-State Network Changes Following Transcranial Magnetic Stimulation in Patients With Aphasia-A Randomized Controlled Study. Neuromodulation. 2022 Jun;25(4):528-537. doi: 10.1016/j.neurom.2021.10.004. Epub 2021 Dec 18. PMID 35088736